CLINICAL TRIAL: NCT05155150
Title: Improving Shared-Decision Making in the Intensive Care Unit Using Patient-reported Outcome Information
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Radboud University Medical Center (Other)
Collaborators: Jeroen Bosch Ziekenhuis (Other)
Responsible Party: Principal Investigator, Marieke Zegers, PhD and Principal Investigator, Radboud University Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 112002
Record Dates: First submitted 2021-11-17; First posted 2021-12-13 (Actual); Last update posted 2023-04-10 (Actual); Status verified 2023-04

CONDITIONS: Intensive Care Unit Syndrome; Patient Engagement
Keywords: Share decision making; Intensive Care Unit; Quality of life
MeSH Terms: conditions — Patient Participation

STUDY DESIGN:
Intervention Model Description: Randomized trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): Providing patient-reported outcome: patients receive personalized information on expected quality of life one year after ICU during ICU admission (during a family meeting)
  Interventions: Behavioral: Providing patient-reported outcome
- Control group (No Intervention): Family meetings take place as usual.

INTERVENTIONS:
Behavioral: Providing patient-reported outcome — Patients receive personalized information on expected quality of life one year after ICU during ICU admission (during a family meeting)
  Arms: Intervention group

SUMMARY:
The aim of this study is to evaluate the effect of incorporation of outcome information in the Intensive Care Unit (ICU) decision-making process on patient and family reported outcomes and experiences of patients, relatives and ICU clinicians in a randomized clinical trial design in the Jeroen Bosch Ziekenhuis and Radboudumc in the Netherlands.

DETAILED DESCRIPTION:
Background Due to advances in critical care medicine, more patients survive their critical illness. However, many Intensive Care Unit (ICU) survivors suffer from physical, cognitive and/or mental problems impacting patients' quality of life (QoL). Because of a lack of long-term outcome information, ICU physicians make decisions regarding ICU treatment based on their clinical experience and intuition. Moreover, patients and relatives are often not involved in the decision-making process.

To improve the ICU decision-making process and to make it more substantiated, the use of patient-reported outcome measures (PROMs) is of utmost importance. Therefore, the Radboudumc, in collaboration with six regional hospitals, including Jeroen Bosch Ziekenhuis (JBZ), set up a large-scale prospective cohort study, MONITOR-IC (www.monitor-ic.nl), to study long-term outcomes of ICU survivors', their QoL and their needs.

This research sets out to evaluate the effect of incorporation of outcome information in the ICU decision-making process on patient and family reported outcomes and experiences of patients, relatives and ICU clinicians in a randomized clinical trial design in the Jeroen Bosch Ziekenhuis and Radboudumc in the Netherlands.

Methods A prediction model for long-term QoL was previously developed using physiological, pathological, drug and treatment data from patients' electronic health record combined with PROMs from one centre of the MONITOR-IC. It was externally validated with the data of six other centres and an E-health tool was developed, incorporating this prediction model. For this research, the E-health tool will be incorporated in family meetings.

ELIGIBILITY:
Inclusion Criteria:

* Patients admitted to the ICU for 12 hours or more
* Patients (or their legal representative) provide written informed consent

Exclusion Criteria:

* Patients admitted to the ICU due to a COVID-19 infection
* Moribund patients

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 160 (Estimated)
Dates: Start 2021-11-09 (Actual); Primary Completion 2023-05 (Estimated); Study Completion 2024-05 (Estimated)

PRIMARY OUTCOMES:
Patient reported experience measure (PREM) | Within 3 months of family meeting
  Patient and/or relative's experience (measured using the CollaboRATE)

SECONDARY OUTCOMES:
Patient reported outcome measure (PROM) | After 3 months and after 1 year
  Quality of life, measured using the EuroQol five-dimensional questionnaire (EQ-5D-5L). The Dutch EQ-5D-5L index ranges from -0.446 to 1, with a higher score indicating a better health related quality of life.
ICU professionals' experiences | Two months before inclusion first patient and two months after inclusion last patient
  Measured using the Ethical Decision-Making Climate Questionnaire (EDMCQ). The EDMCQ consists of three parts: interdisciplinary collaboration and communication (5-point Likert Scale ranging from strongly disagree to strongly agree), leadership by physicians (5-point Likert Scale ranging from never to always) and ethical environment (4-point Likert Scale ranging from strongly disagree to strongly agree). These three parts cover a total of seven factors. Factor scores range from 1-5 or 1-4, with higher scores reflecting more positive views.
Patient reported outcome measure (PROM) | After 3 months and after 1 year
  Anxiety and depression, measured using the Hospital Anxiety and Depression Scale (HADS). The HADS consists of two components (anxiety and depression), with each score ranging from 0-21. A higher score indicates more severe symptoms.

CONTACTS AND LOCATIONS:
Overall Officials: Marieke Zegers, PhD, Principal Investigator — Intensive Care, Radboud university medical center; Koen Simons, MD, PhD, Principal Investigator — Intensive Care, Jeroen Bosch Ziekenhuis; Mark Van den Boogaard, PhD, Principal Investigator — Intensive Care, Radboud university medical center
Locations (2):
- Netherlands (2):
  - Radboud university medical centre, Nijmegen, Gelderland
  - Jeroen Bosch Ziekenhuis, 's-Hertogenbosch, North Brabant

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Porter LL, Simons KS, van der Hoeven JG, van den Boogaard M, Zegers M. Discussing expected long-term quality of life in the ICU: effect on experiences and outcomes of patients, family, and clinicians-a randomized clinical trial. Intensive Care Med. 2025 Mar;51(3):478-489. doi: 10.1007/s00134-025-07812-5. Epub 2025 Feb 24. PMID 39992444